CLINICAL TRIAL: NCT02696785
Title: A Multicenter, Randomized, Double-Blind, Active and Placebo-Controlled 16-Week Study Followed by Long-Term Evaluation of Efficacy and Safety of Ixekizumab (LY2439821) in bDMARD-Naive Patients With Radiographic Axial Spondyloarthritis
Brief Title: A Study of Ixekizumab (LY2439821) in bDMARD-Naive Participants With Radiographic Axial Spondyloarthritis
Acronym: COAST-V
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16178; I1F-MC-RHBV (Other: Eli Lilly and Company); 2015-003932-11 (EudraCT Number)
Record Dates: First submitted 2016-02-26; First posted 2016-03-02 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2018-11

CONDITIONS: Spondyloarthritis
Keywords: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylarthritis; Spondylitis, Ankylosing | interventions — ixekizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Q2W Ixekizumab (Experimental): Double Blind Period: Starting dose of 80 or 160 milligrams (mg) ixekizumab given subcutaneously (SC) at baseline followed by 80 mg ixekizumab given SC every two weeks (Q2W) to week 14.
  Extended Treatment Period: 80 mg ixekizumab given SC Q2W from week 16 to week 52.
  Interventions: Drug: Ixekizumab
- Q4W Ixekizumab (Experimental): Double Blind Period: Starting dose of 80 or 160 mg ixekizumab given SC at baseline followed by 80 mg ixekizumab given SC every four weeks (Q4W) to week 14.
  Extended Treatment Period: 80 mg ixekizumab given SC Q4W from week 16 to week 52.
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator): Double Blind Period: Placebo given SC Q2W to week 14.
  Extended Treatment Period: 80 mg ixekizumab given SC Q2W or Q4W from week 16 to week 52.
  Interventions: Drug: Ixekizumab; Drug: Placebo
- Adalimumab (Active Comparator): Double Blind Period: 40 mg Adalimumab given SC Q2W to week 14.
  Extended Treatment Period: 80 mg ixekizumab given SC Q2W or Q4W from week 20 to week 52.
  Interventions: Drug: Ixekizumab; Drug: Adalimumab

INTERVENTIONS:
Drug: Ixekizumab — Administered SC
  Other Names: LY2439821
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Adalimumab — Administered SC
  Arms: Adalimumab

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of the study drug known as ixekizumab in biological disease-modifying anti-rheumatic drugs (bDMARDs)-naive participants with radiographic axial spondyloarthritis (rad-axSpA).

ELIGIBILITY:
Inclusion Criteria:

* Are ambulatory.
* Diagnosis of radiographic axial spondyloarthritis (rad-xSpA) with sacroiliitis defined radiographically according to the modified New York criteria.
* Participants have a history of back pain ≥3 months with age at onset <45 years.
* In the past had an inadequate response to at least 2 non-steroidal anti-inflammatory drugs (for duration 4 weeks) or cannot tolerate NSAIDS.
* If taking NSAIDS be on a stable dose for at least 2 weeks prior to randomization.
* Have a history of prior therapy for axSpa for at least 12 weeks prior to screening.

Exclusion Criteria:

* Have total ankylosis of the spine.
* Have received any prior, or are currently receiving, treatment with biologics, tumor necrosis factor inhibitors or other immunomodulatory agents.
* Have recently received a live vaccine within 12 weeks or have had a vaccination with Bacillus Calmette-Guerin (BCG) within the past year.
* Have an ongoing or serious infection within the last 12 weeks or evidence of active tuberculosis.
* Have a compromised immune system.
* Have any other serious and/or uncontrolled diseases.
* Have either a current diagnosis or a recent history of malignant disease.
* Have had major surgery within 8 weeks of baseline, or will require surgery during the study.
* Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (19):
  - Arizona Arthritis Research, PLC, Phoenix, Arizona
  - Care Access Research - Huntington Beach, Huntington Beach, California
  - Desert Medical Advances, Palm Desert, California
  - Arthritis Assoc. & Osteoporosis Ctr of Colorado Springs, LLC, Colorado Springs, Colorado
  - Denver Arthritis Center, Denver, Colorado
  - New England Research Associates, Trumbull, Connecticut
  - Sarasota Arthritis Center, Sarasota, Florida
  - Marietta Rheumatology, Marietta, Georgia
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - Klein and Associates MD, PA, Cumberland, Maryland
  - Klein and Associates MD, PA, Hagerstown, Maryland
  - Arthritis Consultants, St Louis, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Shanahan Rheumatology & Immunotherapy, Raleigh, North Carolina
  - Articularis Healthcare Group, INC dba Columbia Arthritis Ctr, Columbia, South Carolina
  - Low Country Research Center, North Charleston, South Carolina
  - Univ of Texas Health Science Center - Houston, Houston, Texas
  - Arthritis Northwest Rheumatology, Spokane, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno, Czechia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin, Germany
- "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Hyōgo, Japan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warszawa, Netherlands
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangjin-gu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Reveille JD, Rudwaleit M, Rahman P, Maldonado-Cocco JA, Magrey M, Bolce R, Ng KJ, Gibble TH, Lisse J, Park SY, Kronbergs A, Navarro-Compan V. Does HLA-B27 Status Influence Ixekizumab Efficacy in Axial Spondyloarthritis? Results From the COAST-V, COAST-W, and COAST-X Trials. Rheumatol Ther. 2026 Feb;13(1):279-291. doi: 10.1007/s40744-025-00810-5. Epub 2025 Dec 19. PMID 41417207
- [Derived] Navarro-Compan V, Reveille JD, Rahman P, Maldonado-Cocco JA, Magrey M, Bolce R, Panni T, Kronbergs A, Rudwaleit M. Ixekizumab Improves Signs, Symptoms, and Quality of Life in Patients with Axial Spondyloarthritis Irrespective of Symptom Duration. Adv Ther. 2025 Sep;42(9):4706-4716. doi: 10.1007/s12325-025-03305-5. Epub 2025 Jul 22. PMID 40694276
- [Derived] Maksymowych WP, Lambert RGW, Bolce RJ, Bello N, Zhu B, Lisse JR, Ostergaard M. The effect of ixekizumab treatment on MRI sacroiliac joint structural lesions in patients with radiographic axial spondyloarthritis: post-hoc analysis of a 52-week, randomised, placebo-controlled trial with an active reference arm. Lancet Rheumatol. 2025 May;7(5):e314-e322. doi: 10.1016/S2665-9913(24)00312-6. Epub 2025 Feb 18. PMID 39983751
- [Derived] Ramiro S, Lukas C, Nissen MJ, Zhu B, Ng KJ, Sheesh M, Doridot G, Liu-Leage S, Chan A, Fang Y, Wei JC. Improvement in spinal pain at night and its impact on long-term outcomes in radiographic axial spondyloarthritis: Results from Ixekizumab COAST-V randomised trial. Semin Arthritis Rheum. 2024 Dec;69:152571. doi: 10.1016/j.semarthrit.2024.152571. Epub 2024 Oct 23. PMID 39509838
- [Derived] Ramiro S, Lukas C, Bessette L, Wickersham P, Panni T, Bolce R, Liu-Leage S, Janos B, Nissen MJ, Wei JC. Early clinical response associates with long-term outcomes with ixekizumab in radiographic axial spondyloarthritis. RMD Open. 2024 Jul 14;10(3):e004429. doi: 10.1136/rmdopen-2024-004429. PMID 39004432
- [Derived] de Vlam K, Maksymowych WP, Gallo G, Rahman P, Mease P, Krishnan V, McVeigh CJ, Lisse J, Zhu D, Bolce RJ, Conaghan PG. Exploring the Effects of Ixekizumab on Pain in Patients with Ankylosing Spondylitis Based on Objective Measures of Inflammation: Post Hoc Analysis from a Large Randomized Clinical Trial. Rheumatol Ther. 2024 Jun;11(3):691-707. doi: 10.1007/s40744-024-00660-7. Epub 2024 Apr 18. PMID 38637464
- [Derived] Deodhar A, Poddubnyy D, Rahman P, Ermann J, Tomita T, Bolce R, Leage SL, Kronbergs A, Johnson C, Araujo J, Leung A, van der Heijde D. Long-Term Safety and Efficacy of Ixekizumab in Patients With Axial Spondyloarthritis: 3-year Data From the COAST Program. J Rheumatol. 2023 Aug;50(8):1020-1028. doi: 10.3899/jrheum.221022. Epub 2023 Feb 15. PMID 36792107
- [Derived] Ortolan A, Ramiro S, Ramonda R, van der Heijde D. External validation of the alternative Ankylosing Spondylitis Disease Activity Score in three randomized clinical trials of ixekizumab. Rheumatology (Oxford). 2023 Jun 1;62(6):2257-2261. doi: 10.1093/rheumatology/keac618. PMID 36282526
- [Derived] van der Horst-Bruinsma IE, de Vlam K, Walsh JA, Bolce R, Hunter T, Sandoval D, Zhu D, Geneus V, Soriano ER, Magrey M. Baseline Characteristics and Treatment Response to Ixekizumab Categorised by Sex in Radiographic and Non-radiographic Axial Spondylarthritis Through 52 Weeks: Data from Three Phase III Randomised Controlled Trials. Adv Ther. 2022 Jun;39(6):2806-2819. doi: 10.1007/s12325-022-02132-2. Epub 2022 Apr 16. PMID 35429281
- [Derived] Maksymowych WP, Bolce R, Gallo G, Seem E, Geneus VJ, Sandoval DM, Ostergaard M, Tada K, Baraliakos X, Deodhar A, Gensler LS. Ixekizumab in radiographic axial spondyloarthritis with and without elevated C-reactive protein or positive magnetic resonance imaging. Rheumatology (Oxford). 2022 Nov 2;61(11):4324-4334. doi: 10.1093/rheumatology/keac104. PMID 35188180
- [Derived] van der Heijde D, Ostergaard M, Reveille JD, Baraliakos X, Kronbergs A, Sandoval DM, Li X, Carlier H, Adams DH, Maksymowych WP. Spinal Radiographic Progression and Predictors of Progression in Patients With Radiographic Axial Spondyloarthritis Receiving Ixekizumab Over 2 Years. J Rheumatol. 2022 Mar;49(3):265-273. doi: 10.3899/jrheum.210471. Epub 2021 Dec 1. PMID 34853086
- [Derived] Deodhar AA, Mease PJ, Rahman P, Navarro-Compan V, Strand V, Hunter T, Bolce R, Leon L, Lauzon S, Marzo-Ortega H. Ixekizumab improves spinal pain, function, fatigue, stiffness, and sleep in radiographic axial Spondyloarthritis: COAST-V/W 52-week results. BMC Rheumatol. 2021 Sep 20;5(1):35. doi: 10.1186/s41927-021-00205-3. PMID 34538257
- [Derived] Dougados M, Wei JC, Landewe R, Sieper J, Baraliakos X, Van den Bosch F, Maksymowych WP, Ermann J, Walsh JA, Tomita T, Deodhar A, van der Heijde D, Li X, Zhao F, Bertram CC, Gallo G, Carlier H, Gensler LS; COAST-V and COAST-W Study Groups. Efficacy and safety of ixekizumab through 52 weeks in two phase 3, randomised, controlled clinical trials in patients with active radiographic axial spondyloarthritis (COAST-V and COAST-W). Ann Rheum Dis. 2020 Feb;79(2):176-185. doi: 10.1136/annrheumdis-2019-216118. Epub 2019 Nov 4. PMID 31685553
- [Derived] Mease P, Walsh JA, Baraliakos X, Inman R, de Vlam K, Wei JC, Hunter T, Gallo G, Sandoval D, Zhao F, Dong Y, Bolce R, Marzo-Ortega H. Translating Improvements with Ixekizumab in Clinical Trial Outcomes into Clinical Practice: ASAS40, Pain, Fatigue, and Sleep in Ankylosing Spondylitis. Rheumatol Ther. 2019 Sep;6(3):435-450. doi: 10.1007/s40744-019-0165-3. Epub 2019 Jun 28. PMID 31254223
- See also: Click here for more information about this study: A Study of Ixekizumab (LY2439821) in bDMARD-Naive Participants With Radiographic Axial Spondyloarthritis (COAST-V) — http://www.lillytrialguide.com/en-US/studies/axial-spondyloarthritis%20(ankylosing%20spondylitis)/RHBV#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Blinded treatment period (Week 0 to Week 16), followed by extended treatment period (Week 16 to Week 52), followed by post treatment period for a maximum of 24 weeks.
  Washout period occurred for only Adalimumab group for 6 weeks (Week 14 to Week 20).
Pre-assignment Details: Participants who completed study were eligible to enroll into a long-term study (Study I1F-MC-RHBY [RHBY]) for up to 2 additional years. Participants that do not enroll into study RHBY will complete the Post-Treatment Follow-Up Period.
Groups:
- PBO/IXE: Blinded Treatment Period: Participants received placebo every two weeks by subcutaneous injection.
  Extended Treatment Period: Participants received starting dose of 160mg Ixekizumab at week 16 followed by 80mg Ixekizumab either every two weeks (Q2W) or every four weeks (Q4W) by subcutaneous (SC) injection during extended treatment period.
  Participants did not receive any intervention during Follow-up period.
- ADA/PBO/IXE: Blinded Treatment Period:Participants received 40mg Adalimumab every two weeks by SC injection.
  Washout Period: Participants received placebo for 6 weeks. Extended Treatment Period:Participants received 80mg Ixekizumab either Q2W or Q4W by SC injection during extension treatment period.
  Participants did not receive any intervention during Follow-up period.
- IXE80Q2W/IXE80Q2W: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every two weeks by subcutaneous injection during blinded & extension treatment period.
  Participants did not receive any intervention during Follow-up period.
- IXE80Q4W/IXE80Q4W: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every four weeks by subcutaneous injection during blinded & extension treatment period.
  Participants did not receive any intervention during Follow-up period.
Period: Blinded Treatment Period
Arm/Group | PBO/IXE | ADA/PBO/IXE | IXE80Q2W/IXE80Q2W | IXE80Q4W/IXE80Q4W
Started | 87 | 90 | 83 | 81
Received at Least One Dose of Study Drug | 86 | 90 | 83 | 81
Completed | 86 | 88 | 79 | 78
Not Completed | 1 | 2 | 4 | 3
Not completed — Adverse Event | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Screen Failure | 1 | 0 | 0 | 0
Period: Washout Period
Arm/Group | PBO/IXE | ADA/PBO/IXE | IXE80Q2W/IXE80Q2W | IXE80Q4W/IXE80Q4W
Started | 0 (Washout period occurred only for Adalimumab group.) | 88 | 0 (Washout period occurred only for Adalimumab group.) | 0 (Washout period occurred only for Adalimumab group.)
Completed | 0 | 86 | 0 | 0
Not Completed | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Period: Extended Treatment Period
Arm/Group | PBO/IXE | ADA/PBO/IXE | IXE80Q2W/IXE80Q2W | IXE80Q4W/IXE80Q4W
Started | 86 | 86 | 79 | 78
Completed | 83 | 80 | 74 | 72
Not Completed | 3 | 6 | 5 | 6
Not completed — Adverse Event | 2 | 3 | 2 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 3 | 5
Period: Follow-up Period
Arm/Group | PBO/IXE | ADA/PBO/IXE | IXE80Q2W/IXE80Q2W | IXE80Q4W/IXE80Q4W
Started | 1 (Participants who completed study were eligible to enroll RHBY & who didn't enroll entered Follow-Up.) | 0 (Participants who completed study were eligible to enroll RHBY & who didn't enroll entered Follow-Up.) | 24 (Participants who completed study were eligible to enroll RHBY & who didn't enroll entered Follow-Up.) | 16 (Participants who completed study were eligible to enroll RHBY & who didn't enroll entered Follow-Up.)
Completed | 0 | 0 | 11 | 8
Not Completed | 1 | 0 | 13 | 8
Not completed — Adverse Event | 0 | 0 | 8 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 5 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- PBO/IXE: Participants received placebo every two weeks by subcutaneous injection during blinded treatment period and 80mg Ixekizumab either Q2W or Q4W by subcutaneous injection during extension treatment period.
- ADA/IXE: Participants received 40mg Adalimumab every two weeks by SC injection during blinded treatment period and 80mg Ixekizumab either Q2W or Q4W by SC injection during extension treatment period.
- IXE80Q2W/IXE80Q2W: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every two weeks by subcutaneous injection during blinded & extension treatment period.
- IXE80Q4W/IXE80Q4W: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every four weeks by subcutaneous injection during blinded & extension treatment period.
- Total: Total of all reporting groups
Arm/Group | PBO/IXE | ADA/IXE | IXE80Q2W/IXE80Q2W | IXE80Q4W/IXE80Q4W | Total
Number analyzed (Participants) | 86 | 90 | 83 | 81 | 340
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (12.01) | 41.8 (11.44) | 41.3 (11.17) | 41.0 (12.13) | 41.7 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 19 | 13 | 64
  Male | 71 | 73 | 64 | 68 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 8 | 8 | 34
  Not Hispanic or Latino | 67 | 74 | 68 | 66 | 275
  Unknown or Not Reported | 8 | 9 | 7 | 7 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 4 | 4 | 14
  Asian | 28 | 29 | 25 | 25 | 107
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 52 | 57 | 52 | 52 | 213
  More than one race | 2 | 2 | 2 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 10 | 14 | 12 | 11 | 47
  Netherlands | 0 | 2 | 2 | 0 | 4
  United States | 5 | 3 | 4 | 3 | 15
  Czechia | 14 | 14 | 13 | 13 | 54
  Japan | 3 | 3 | 0 | 1 | 7
  Taiwan | 13 | 12 | 13 | 13 | 51
  Germany | 0 | 2 | 1 | 0 | 3
  Canada | 2 | 3 | 2 | 2 | 9
  Hungary | 3 | 2 | 2 | 3 | 10
  Mexico | 8 | 7 | 8 | 7 | 30
  Poland | 16 | 15 | 15 | 16 | 62
  Russia | 12 | 13 | 11 | 12 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Assessment of Spondyloarthritis International Society 40 (ASAS40) Response
Description: ASAS40 is defined as improvement from baseline of greater than or equal to (>=) 40% and absolute improvement from baseline of at least 2 units in at least 3 of the following 4 domains without any worsening in the remaining domains.
  1. Patient Global: How active was your spondylitis on average during the last week? score range 0 (not active) to 10 (very active).
  2. Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  3. Bath Ankylosing Spondylitis Functional Index: Participant is asked to rate the difficulty associated with 10 individual basic functional activities. Participants response is captured using numeric rating scale (NRS) scale (range 0 to 10) with a higher score indicating worse function.
  4. Inflammation based on Q5 & Q6 mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe).
Time Frame: Week 16
Population: All Randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo every two weeks by subcutaneous injection.
- Adalimumab: Participants received 40mg Adalimumab every two weeks by SC injection.
- IXE80Q4W: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every four weeks by subcutaneous injection.
- IXE80Q2W: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every two weeks by subcutaneous injection.
Arm/Group | Placebo | Adalimumab | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
percentage of participants | 18.4 | 35.6 | 48.1 | 51.8
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; Overall Work Impairment Score; Test type: Superiority; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 2.73, 95% CI 2-sided [1.35 to 5.52]
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Overall Work Impairment Score; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.45, 95% CI 2-sided [2.20 to 9.03]
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Overall Work Impairment Score; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.09, 95% CI 2-sided [2.52 to 10.28]
Statistical Analysis 4: Comparison: Placebo vs Adalimumab; Percentage of Activity Impairment; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -7.0, 95% CI 2-sided [-13.2 to -0.7], Standard Error of Mean 3.16
Statistical Analysis 5: Comparison: Placebo vs IXE80Q2W; Percentage of Activity Impairment; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -9.3, 95% CI 2-sided [-15.5 to -3.0], Standard Error of Mean 3.19
Statistical Analysis 6: Comparison: Placebo vs IXE80Q4W; Percentage of Activity Impairment; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -8.9, 95% CI 2-sided [-15.2 to -2.5], Standard Error of Mean 3.22

2. Secondary Outcome: Percentage of Participants Achieving an ASAS20 Response
Description: ASAS20 response is defined as a ≥20% improvement and an absolute improvement from baseline of ≥1 units in ≥3 of 4 following domains and no worsening of ≥20% and ≥1 unit (range 0 to 10) in the remaining domain.
  1. Patient Global: How active was your spondylitis on average during the last week? score range 0 (not active) to 10 (very active).
  2. Spinal Pain: How much Pain of your spine due to Ankylosing spondylitis? score ranges 0 (no pain) to 10 (severe pain).
  3. Bath Ankylosing Spondylitis Functional Index: Participant is asked to rate the difficulty associated with 10 individual basic functional activities. Participants response is captured using NRS scale (range 0 to 10) with a higher score indicating worse function.
  4. Inflammation based on Q5 & Q6 mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (mean of intensity & duration of stiffness): Score ranges from "0" (none) and "10" (very severe).
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Groups:
- Adalimumab 40mg: Participants received 40mg Adalimumab every two weeks by SC injection.
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
percentage of participants | 40.2 | 58.9 | 64.2 | 68.7
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.25 to 4.23]
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.48 to 5.24]
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.39, 95% CI 2-sided [1.79 to 6.41]

3. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS)
Description: ASDAS is a composite index to assess disease activity in AS. The parameters used for the ASDAS (with CRP as acute phase reactant) are the following:
  1. Total back pain
  2. Patient global
  3. Peripheral pain/swelling
  4. Duration of morning stiffness
  5. CRP in mg/L The ASDAScrp is calculated with the following equation: 0.121 × total back pain + 0.110 × patient global + 0.073 × peripheral pain/swelling + 0.058 × duration of morning stiffness + 0.579 × Ln(CRP+1). CRP is in mg/liter, the range of other variables is from 0 to 10.Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher scores indicated higher disease activity. Ln represents the natural logarithm.
  Least Square (LS) Mean was calculated using mixed model repeated measures (MMRM) model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
score on a scale | -0.46 (0.099) | -1.30 (0.096) | -1.43 (0.102) | -1.37 (0.101)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.84, 95% CI 2-sided [-1.11 to -0.57], Standard Error of Mean 0.137
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.97, 95% CI 2-sided [-1.25 to -0.70], Standard Error of Mean 0.141
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.91, 95% CI 2-sided [-1.18 to -0.63], Standard Error of Mean 0.140

4. Secondary Outcome: Percentage of Participants Achieving Bath Ankylosing Spondylitis Disease Activity Index 50 (BASDAI50) Response
Description: The BASDAI is a participant-reported assessment consisting of 6 questions that relate to 5 major symptoms relevant to radiographic axial spondyloarthritis measuring discomfort, pain, and fatigue. 1) Fatigue, 2) Spinal pain, 3) Peripheral arthritis, 4) Enthesitis, 5) Intensity, and 6) Duration of morning stiffness. participants need to score each item with a score from 0 to 10 (NRS). total score is obtained from the average of symptom scores ranging 0 (no problem) to 10 (worst problem).
  BASDAI50 represents an improvement of ≥50% of the BASDAI score from baseline.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
percentage of participants | 17.2 | 32.2 | 42.0 | 43.4
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.23 to 5.21]
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.74, 95% CI 2-sided [1.82 to 7.70]
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.90, 95% CI 2-sided [1.91 to 7.98]

5. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The BASFI is a participant-reported assessment that establishes a participants functional baseline and subsequent response to treatment. To complete the BASFI, a participant is asked to rate the difficulty associated with 10 individual basic functional activities. Participants respond to each question using an NRS scale (range 0 to 10) with a higher score indicating worse function. The participants final BASFI score is the mean of the 10 item scores has a possible minimum value of 0 and a possible maximum value of 10, with a higher score indicating worse function.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
score on a scale | -1.16 (0.215) | -2.14 (0.209) | -2.39 (0.222) | -2.43 (0.219)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean Difference = -0.97, 95% CI 2-sided [-1.56 to -0.39], Standard Error of Mean 0.299
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.22, 95% CI 2-sided [-1.83 to -0.62], Standard Error of Mean 0.307
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.27, 95% CI 2-sided [-1.86 to -0.67], Standard Error of Mean 0.304

6. Secondary Outcome: Percentage of Participants Achieving ASDAS Inactive Disease
Description: ASDAS is a composite index to assess disease activity in AS. The parameters used for the ASDAS (with CRP as acute phase reactant) are the following:
  1. Total back pain
  2. Patient global
  3. Peripheral pain/swelling
  4. Duration of morning stiffness
  5. CRP in mg/L The ASDAScrp is calculated with the following equation: 0.121 × total back pain + 0.110 × patient global + 0.073 × peripheral pain/swelling + 0.058 × duration of morning stiffness + 0.579 × Ln(CRP+1). CRP is in mg/liter, the range of other variables is from 0 to 10.Data from five variables combined to yield a score (0.6361 to no defined upper limit), where higher scores indicated higher disease activity. Ln represents the natural logarithm. ASDAS Inactive Disease is defined as a score of <1.3.
Time Frame: Week 16
Population: All randomized participants.
Measure: Number; unit: percentage of Participants
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
percentage of Participants | 2.3 | 15.6 | 16.0 | 10.8
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.009, Regression, Logistic; LSMean Difference = 7.62, 95% CI 2-sided [1.67 to 34.68]
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.007, Regression, Logistic; Odds Ratio (OR) = 8.03, 95% CI 2-sided [1.75 to 36.83]
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.041, Regression, Logistic; Odds Ratio (OR) = 5.13, 95% CI 2-sided [1.07 to 24.49]

7. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Ankylosing Spondylitis Spinal Magnetic Resonance Imaging [ASSpiMRI] - Berlin Score)
Description: The Berlin modification of Ankylosing Spondylitis spine MRI score for activity (ASspiMRI) scoring technique assesses inflammation in each of 23 disco-vertebral units (DVU). All 23 disco-vertebral units (DVU) of the spine (from C2 to S1) are scored for bone marrow edema. Scores for each DVU range from 0-3 (0=normal; 1=minor bone marrow edema [less than or equal to 25% of DVU; 3=severe bone marrow edema (more that 50% of DVU)]. The composite score ranges from 0 to 69, with higher scores reflecting worse disease.
  Least Squares (LS) Mean was calculated using ANCOVA model with treatment, geographic region, baseline CRP status and baseline value as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and week 16 Berlin score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 81 | 82 | 78 | 76
score on a scale | -0.15 (0.323) | -2.92 (0.314) | -2.77 (0.328) | -2.54 (0.330)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -2.78, 95% CI 2-sided [-3.7 to -1.9], Standard Error of Mean 0.447
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -2.62, 95% CI 2-sided [-3.5 to -1.7], Standard Error of Mean 0.450
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -2.39, 95% CI 2-sided [-3.3 to -1.5], Standard Error of Mean 0.452

8. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: The SF-36 is a 36-item participant administered measure designed to be a short, multipurpose assessment of health in the areas of physical functioning, role - physical, role - emotional, bodily pain, vitality, social functioning, mental health, and general health. The 2 overarching domains of mental well- being and physical well-being are captured by the Mental Component Summary and Physical Component Summary scores. T-scores are used for analysis. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
score on a scale
  PCS | 3.6432 (0.7530) | 6.9005 (0.7310) | 7.6952 (0.7768) | 7.9686 (0.7665)
  MCS | 2.1229 (0.8431) | 2.5550 (0.8225) | 2.7502 (0.8763) | 2.5696 (0.8650)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; PCS; Test type: Superiority; p = 0.002, Mixed Models Analysis; LSMean Difference = 3.2574, 95% CI 2-sided [1.2041 to 5.3106], Standard Error of Mean 1.0437
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; PCS; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 4.0520, 95% CI 2-sided [1.9432 to 6.1608], Standard Error of Mean 1.0720
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; PCS; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = 4.3254, 95% CI 2-sided [2.2321 to 6.4186], Standard Error of Mean 1.0641
Statistical Analysis 4: Comparison: Placebo vs Adalimumab 40mg; MCS; Test type: Superiority; p = 0.713, Mixed Models Analysis; LSMean Difference = 0.4321, 95% CI 2-sided [-1.8732 to 2.7373], Standard Error of Mean 1.1718
Statistical Analysis 5: Comparison: Placebo vs IXE80Q4W; MCS; Test type: Superiority; p = 0.602, Mixed Models Analysis; LSMean Difference = 0.6273, 95% CI 2-sided [-1.7387 to 2.9934], Standard Error of Mean 1.2028
Statistical Analysis 6: Comparison: Placebo vs IXE80Q2W; MCS; Test type: Superiority; p = 0.709, Mixed Models Analysis; LSMean Difference = 0.4467, 95% CI 2-sided [-1.9097 to 2.8030], Standard Error of Mean 1.1978

9. Secondary Outcome: Change From Baseline in ASAS Health Index (ASAS HI)
Description: ASAS HI is a disease-specific health-index instrument designed to assess the impact of interventions for SpA, including axSpA. The 17-item instrument has scores ranging from 0 (good health) to 17 (poor health). Each item consists of one question that the participant needs to respond to with either "I agree" (score of 1) or "I do not agree" (score of 0). A score of "1" is given where the item is affirmed, indicating adverse health. All item scores are summed to give a total score or index.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
score on a scale | -1.25 (0.300) | -2.30 (0.292) | -2.36 (0.311) | -2.74 (0.306)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.012, Mixed Models Analysis; LSMean Difference = -1.05, 95% CI 2-sided [-1.87 to -0.23], Standard Error of Mean 0.416
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.010, Mixed Models Analysis; LSMean Difference = -1.11, 95% CI 2-sided [-1.95 to -0.27], Standard Error of Mean 0.428
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -1.49, 95% CI 2-sided [-2.32 to -0.66], Standard Error of Mean 0.423

10. Secondary Outcome: Change From Baseline in the Measure of High Sensitivity C-Reactive Protein (CRP)
Description: High sensitivity CRP is the measure of acute phase reactant. It will be measured with a high sensitivity assay at the central laboratory to help assess the effect of Ixekizumab on disease activity.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, visit and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Milliragm per Litre (mg/mL)
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
Milliragm per Litre (mg/mL) | 1.426 (1.9244) | -7.202 (1.8688) | -5.209 (1.9803) | -6.565 (1.9582)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean Difference = -8.628, 95% CI 2-sided [-13.885 to -3.371], Standard Error of Mean 2.6724
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.016, Mixed Models Analysis; LSMean Difference = -6.635, 95% CI 2-sided [-12.033 to -1.238], Standard Error of Mean 2.7438
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.004, Mixed Models Analysis; LSMean Difference = -7.991, 95% CI 2-sided [-13.351 to -2.631], Standard Error of Mean 2.7248

11. Secondary Outcome: Change From Baseline in Mobility on the Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: The BASMI is a combined index comprising the following 5 clinical measurements of spinal mobility in participants with rad-axSpA.
  1. Lateral spinal flexion
  2. Tragus-to-wall distance
  3. Lumbar flexion (modified Schrober)
  4. Maximal intermalleolar distance
  5. Cervical rotation. The BASMI includes these 5 measurements that are each scaled to a score of 0 to 10 depending on the result of the assessment (BASMI linear function). The average score of the 5 assessments gives the BASMI linear result. The higher the BASMI score the more severe the participants limitation of movement due to their AS.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
score on a scale | -0.080 (0.0826) | -0.447 (0.0800) | -0.502 (0.0858) | -0.408 (0.0840)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.001, Mixed Models Analysis; LSMean Difference = -0.367, 95% CI 2-sided [-0.592 to -0.142], Standard Error of Mean 0.1143
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -0.422, 95% CI 2-sided [-0.655 to -0.189], Standard Error of Mean 0.1184
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.005, Mixed Models Analysis; LSMean Difference = -0.329, 95% CI 2-sided [-0.558 to -0.099], Standard Error of Mean 0.1167

12. Secondary Outcome: Change From Baseline in Chest Expansion
Description: While participants have their hands resting on or behind the head, the assessor has measured the chest's encircled length by centimeter at the fourth intercostal level anteriorly. The difference between maximal inspiration and expiration in centimeters was recorded. Two tries were recorded. The better measurement (larger difference) of 2 tries (in centimeters) was used for analyses.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All Randomized Participants.
Measure: Least Squares Mean (Standard Error); unit: Centimeters (cm)
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
Centimeters (cm) | 0.06 (0.152) | 0.70 (0.148) | 0.49 (0.158) | 0.67 (0.155)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.003, Mixed Models Analysis; LSMean Difference = 0.63, 95% CI 2-sided [0.22 to 1.05], Standard Error of Mean 0.211
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.051, Mixed Models Analysis; LSMean Difference = 0.43, 95% CI 2-sided [-0.00 to 0.86], Standard Error of Mean 0.219
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.005, Mixed Models Analysis; LSMean Difference = 0.60, 95% CI 2-sided [0.18 to 1.03], Standard Error of Mean 0.215

13. Secondary Outcome: Change From Baseline in Occiput to Wall Distance
Description: The participant is to make a maximum effort to touch the head against the wall when standing with heels and back against the wall (occiput). Then the distance from occiput to wall is measured. Two tries will be recorded. The better (smaller) measurement of 2 tries (in centimeters) will be used for analyses.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
cm | -0.06 (0.232) | -0.72 (0.225) | -0.69 (0.240) | -0.73 (0.236)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.039, Mixed Models Analysis; LSMean Difference = -0.67, 95% CI 2-sided [-1.30 to -0.03], Standard Error of Mean 0.321
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.057, Mixed Models Analysis; LSMean Difference = -0.63, 95% CI 2-sided [-1.28 to 0.02], Standard Error of Mean 0.330
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.042, Mixed Models Analysis; LSMean Difference = -0.67, 95% CI 2-sided [-1.31 to -0.03], Standard Error of Mean 0.327

14. Secondary Outcome: Change From Baseline in MRI Sacroiliac Joint(s) (SIJ) Spondyloarthritis Research Consortium of Canada (SPARCC) Score
Description: Both left and right SIJ are scored for bone marrow edema.Each side has 6 slices and each slice has 6 scoring units, and each scoring unit has a score of 0 or 1. Total SIJ SPARCC scores can range from 0 to 72 with higher scores reflecting worse disease.
  LSMean was calculated using ANCOVA model with treatment, geographic region, baseline CRP status and baseline value as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and week 16 SPARCC score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 81 | 82 | 78 | 77
score on a scale | 0.92 (0.582) | -4.21 (0.568) | -3.97 (0.590) | -4.25 (0.591)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -5.13, 95% CI 2-sided [-6.7 to -3.5], Standard Error of Mean 0.806
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -4.89, 95% CI 2-sided [-6.5 to -3.3], Standard Error of Mean 0.812
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -5.17, 95% CI 2-sided [-6.8 to -3.6], Standard Error of Mean 0.816

15. Secondary Outcome: Change From Baseline in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES)
Description: The MASES is an index used to measure the severity of enthesitis .The MASES assesses 13 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include costochondral 1 (right/left), costochondral 7 (right/left), spinal iliaca anterior superior (right/left), crista iliaca (right/left), spina iliaca posterior (right/left), processus spinosus L5, and Achilles tendon proximal insertion (right/left). The MASES is the sum of all site scores (range 0 to 13); higher scores indicate more severe enthesitis.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline MASES score > 0.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 56 | 51 | 49 | 50
score on a scale | -2.1 (0.34) | -2.6 (0.34) | -2.3 (0.36) | -2.4 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.317, Mixed Models Analysis; LSMean Difference = -0.5, 95% CI 2-sided [-1.4 to 0.5], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.683, Mixed Models Analysis; LSMean Difference = -0.2, 95% CI 2-sided [-1.1 to 0.8], Standard Error of Mean 0.48
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.500, Mixed Models Analysis; LSMean Difference = -0.3, 95% CI 2-sided [-1.3 to 0.6], Standard Error of Mean 0.48

16. Secondary Outcome: Change From Baseline in SPARCC Enthesitis Score
Description: The SPARCC enthesitis is an index used to measure the severity of enthesitis. The SPARCC assesses 16 sites for enthesitis using a score of "0" for no activity or "1" for activity. Sites assessed include Medial epicondyle (left/right [L/R]), Lateral epicondyle (L/R), Supraspinatus insertion into greater tuberosity of humerus (L/R), Greater trochanter (L/R), Quadriceps insertion into superior border of patella (L/R), Patellar ligament insertion into inferior pole of patella or tibial tubercle (L/R), Achilles tendon insertion into calcaneum (L/R), and Plantar fascia insertion into calcaneum (L/R). The SPARCC is the sum of all site scores (range 0 to 16). Higher scores indicate more severe enthesitis.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline SPARCC score > 0.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 41 | 40 | 40 | 35
score on a scale | -2.1 (0.40) | -2.9 (0.40) | -2.7 (0.40) | -2.6 (0.43)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.154, Mixed Models Analysis; LSMean Difference = -0.8, 95% CI 2-sided [-1.9 to 0.3], Standard Error of Mean 0.56
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = -0.6, Mixed Models Analysis; LSMean Difference = 0.255, 95% CI 2-sided [-1.8 to 0.5], Standard Error of Mean 0.56
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.398, Mixed Models Analysis; LSMean Difference = -0.5, 95% CI 2-sided [-1.6 to 0.7], Standard Error of Mean 0.58

17. Secondary Outcome: Change From Baseline in Severity of Peripheral Arthritis by Tender (TJC)
Description: The number of tender and painful joints was determined by examination of 46 joints (23 joints on each side of the participants body. The 46 joints are assessed and classified as tender or not tender. sum of all joints checked to be tender/painful divided by number of evaluable joints which is multiplied by 46 to obtain TJC score. The scores ranges from 0 (no tender/painful joints) to 46 (all joints tender/painful).
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline TJC > 0.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 51 | 49 | 44 | 45
score on a scale | -2.0 (0.53) | -2.2 (0.55) | -2.5 (0.58) | -3.3 (0.58)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.783, Mixed Models Analysis; LSMean Difference = -0.2, 95% CI 2-sided [-1.7 to 1.3], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.550, Mixed Models Analysis; LSMean Difference = -0.5, 95% CI 2-sided [-2.0 to 1.1], Standard Error of Mean 0.78
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.091, Mixed Models Analysis; LSMean Difference = -1.3, 95% CI 2-sided [-2.8 to 0.2], Standard Error of Mean 0.77

18. Secondary Outcome: Number of Participants With Anterior Uveitis or Uveitis Flares
Description: Anterior uveitis is an inflammation of the middle layer of the eye which includes the iris (colored part of the eye) and the adjacent tissue, known as the ciliary body.
Time Frame: Baseline through Week 16
Population: All randomized participants.
Measure: Number; unit: Count of Participants
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
Count of Participants | 0 | 0 | 1 | 0

19. Secondary Outcome: Change From Baseline in the Fatigue Numeric Rating Scale (NRS) Score
Description: The Fatigue Severity NRS is a participant-administered, single-item, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no fatigue" and 10 representing "as bad as you can imagine". Participants rate their fatigue (feeling tired or worn out) by circling the one number that describes their worst level of fatigue during the previous 24 hours.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Participants placebo every two weeks by subcutaneous injection.
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
score on a scale | -1.4 (0.23) | -2.2 (0.23) | -2.5 (0.24) | -2.1 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.027, Mixed Models Analysis; LSMean Difference = -0.7, 95% CI 2-sided [-1.3 to -0.1], Standard Error of Mean 0.32
Statistical Analysis 2: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.002, Mixed Models Analysis; LSMean Difference = -1.0, 95% CI 2-sided [-1.7 to -0.4], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.035, Mixed Models Analysis; LSMean Difference = -0.7, 95% CI 2-sided [-1.3 to -0.0], Standard Error of Mean 0.33

20. Secondary Outcome: Change From Baseline in the Jenkins Sleep Evaluation Questionnaire (JSEQ)
Description: The JSEQ is a 4-item scale designed to estimate sleep problems in clinical research. The JSEQ assesses the frequency of sleep disturbance in 4 categories: 1) trouble falling asleep, 2) waking up several times during the night, 3) having trouble staying asleep (including waking up far too early), and 4) waking up after the usual amount of sleep feeling tired and worn out. Participants report the number of days they experience each of these problems in the past month on a 6-point Likert scale ranging from 0 = "no days" to 5 = "22-30 days." The total JSEQ score ranges from 0 to 20, with higher scores indicating greater sleep disturbance.
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
score on a scale | -1.5 (0.41) | -2.7 (0.40) | -2.5 (0.43) | -3.0 (0.42)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.041, Mixed Models Analysis; LSMean Difference = -1.2, 95% CI 2-sided [-2.3 to -0.0], Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.125, Mixed Models Analysis; LSMean Difference = -0.9, 95% CI 2-sided [-2.1 to 0.3], Standard Error of Mean 0.59
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.013, Mixed Models Analysis; LSMean Difference = -1.4, 95% CI 2-sided [-2.6 to -0.3], Standard Error of Mean 0.58

21. Secondary Outcome: Change From Baseline in the Work Productivity Activity Impairment Spondyloarthritis (WPAI-SpA) Scores
Description: The WPAI-SpA consists of 6 questions to determine employment status, hours missed from work because of SpA, hours missed from work for other reasons, hours actually worked, the degree to which SpA affected work productivity while at work, and the degree to which SpA affected activities outside of work. The WPAI-SpA has been validated in the rad-axSpA patient population. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. The computed percentage range for each sub-scale was from 0-100. Greater scores indicate greater impairment and less productivity.
  LSMean was calculated using ANCOVA model with treatment, geographic region, baseline CRP status and baseline value as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
score on a scale
  Overall Work Impairment Score | -17.82 (3.254) | -21.44 (2.921) | -21.36 (3.061) | -24.06 (3.299)
  Percentage of Activity Impairment | -14.1 (2.28) | -21.1 (2.22) | -23.0 (2.35) | -23.4 (2.30)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.989, Mixed Models Analysis; LSMean Difference = 0.04, 95% CI 2-sided [-6.03 to 6.12], Standard Error of Mean 3.082
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.429, Mixed Models Analysis; LSMean Difference = 2.50, 95% CI 2-sided [-3.71 to 8.70], Standard Error of Mean 3.146
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.096, Mixed Models Analysis; LSMean Difference = -5.47, 95% CI 2-sided [-11.92 to 0.98], Standard Error of Mean 3.270

22. Secondary Outcome: Change From Baseline in ASAS-Nonsteroidal Anti-Inflammatory Drug (NSAID) Score
Description: ASAS-NSAID score is used to present the NSAID intake by considering the type of NSAID, the total dose, & the number of days taking NSAID during a period of interest (PI).. ASAS-NSAID score=(equivalent NSAID score)x(days of intake during PI)x(days per week)/(PI in days). Higher scores indicate greater NSAIDs intake. 0= no intake, 100 = equivalent NSAID intake.
Time Frame: Baseline, Week 52
Population: Participants in Extended Treatment Period Population Who had NSAID Intake at Baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo/Ixekizumab: Participants received placebo every two weeks during blinded treatment period and starting dose of 160mg Ixekizumab at week 16 followed by 80mg Ixekizumab either Q2W or Q4W extended treatment period by subcutaneous injection.
- Adalimumab/Ixekizumab: Participants received 40mg Adalimumab every two weeks during blinded treatment period and 80mg Ixekizumab either Q2W or Q4W during extended treatment period by subcutaneous injection.
- Ixekizumab Q4W/Ixekizumab Q4W; Ixekizumab 80mg Q2W/Ixekizumab 80mg Q2W: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every four weeks during blinded treatment and extension period by subcutaneous injection.
Arm/Group | Placebo/Ixekizumab | Adalimumab/Ixekizumab | Ixekizumab Q4W/Ixekizumab Q4W | Ixekizumab 80mg Q2W/Ixekizumab 80mg Q2W
Number analyzed (Participants) | 78 | 80 | 71 | 76
score on a scale | -10.28 (27.472) | -5.91 (20.861) | -7.62 (25.430) | -9.91 (27.940)

23. Secondary Outcome: Number of Participants With Anti Ixekizumab Antibodies
Description: A treatment emergent - antidrug antibody (TE-ADA) positive patient is defined as: a) a patient with a >= 4-fold increase over a positive baseline antibody titer; or b) for a negative baseline titer, a patient with an increase from the baseline to a level of >= 1:10.
Time Frame: Week 16
Population: All randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 87 | 90 | 81 | 83
Participants | 2 | 5 | 2 | 2

24. Secondary Outcome: Pharmacokinetics: Trough Ixekizumab Concentration at Steady State (Ctrough ss)
Time Frame: Week 16
Population: All randomized participants who received at least one dose of Ixekizumab.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per millilitre (μg/mL)
Groups:
- IXE80Q4W: Participants received 80mg Ixekizumab every four weeks by subcutaneous injection.
- IXE160/80Q4W: Participants received starting dose of 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every four weeks by subcutaneous injection.
- IXE80Q2W: Participants received 80mg Ixekizumab every two weeks by subcutaneous injection.
- IXE160/80Q2W: Participants received starting dose of 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every two weeks by subcutaneous injection.
Arm/Group | IXE80Q4W | IXE160/80Q4W | IXE80Q2W | IXE160/80Q2W
Number analyzed (Participants) | 42 | 39 | 45 | 38
microgram per millilitre (μg/mL) | 3.56 (56) | 3.88 (55) | 11.6 (54) | 11.3 (43)

25. Secondary Outcome: Change From Baseline in Severity of Peripheral Arthritis by Swollen Joint Count (SJC)
Description: The number of swollen joints was determined by examination of 44 joints (22 joints on each side of the participants body. The 44 joints are assessed and classified as swollen or not swollen. "sum of all joints checked to be swollen" divided by "number of evaluable joints" and then multiplied by 44 to obtain SJC score. The SJC score ranges from 0 (no swollen joints) to 44 (all joints swollen).
  LSMean was calculated using MMRM model with treatment, geographic region, baseline CRP status, baseline value, visit, baseline value-by-visit, and treatment-by-visit interaction as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline SJC > 0.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab 40mg | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 22 | 23 | 24 | 22
score on a scale | -1.7 (0.55) | -2.7 (0.53) | -3.6 (0.53) | -2.7 (0.57)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40mg; Test type: Superiority; p = 0.166, Mixed Models Analysis; LSMean Difference = -1.1, 95% CI 2-sided [-2.6 to 0.4], Standard Error of Mean 0.76
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p = 0.011, Mixed Models Analysis; LSMean Difference = -1.9, 95% CI 2-sided [-3.4 to -0.4], Standard Error of Mean 0.73
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p = 0.182, Mixed Models Analysis; LSMean Difference = -1.0, 95% CI 2-sided [-2.6 to 0.5], Standard Error of Mean 0.77

26. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging (MRI) of the Spine (Spondyloarthritis Research Consortium of Canada [SPARCC] Score)
Description: MRI score of spine was assessed using SPARCC method. All 23 disco-vertebral units (DVUs) of the spine (from C2 to S1) are scored for bone marrow edema. A single DVU has a scoring range of 0 to 18, bringing the maximum total score to 414, with higher scores reflecting worse disease. Scoring was performed by central readers.
  LSMean was calculated using ANCOVA model with treatment, geographic region, baseline CRP status and baseline value as fixed factors
Time Frame: Baseline, Week 16
Population: All randomized participants with baseline and week 16 SPARCC MRI score for spine.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Adalimumab | IXE80Q4W | IXE80Q2W
Number analyzed (Participants) | 81 | 82 | 78 | 76
score on a scale | -1.51 (1.147) | -11.57 (1.113) | -11.02 (1.160) | -9.58 (1.168)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -10.07, 95% CI 2-sided [-13.2 to -6.9], Standard Error of Mean 1.588
Statistical Analysis 2: Comparison: Placebo vs IXE80Q4W; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -9.51, 95% CI 2-sided [-12.6 to -6.4], Standard Error of Mean 1.591
Statistical Analysis 3: Comparison: Placebo vs IXE80Q2W; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference = -8.08, 95% CI 2-sided [-11.2 to -4.9], Standard Error of Mean 1.603

ADVERSE EVENTS:
Time Frame: Upto 76 Weeks
Description: All randomized participants who received at least one dose of study drug. There are gender specific adverse events, only occurring in male or female participants. The number of participants exposed has been adjusted accordingly.
Groups:
- Placebo - Blinded Treatment: Participants received placebo every two weeks by subcutaneous injection.
- Adalimumab 40mg - Blinded Treatment: Participants received 40mg Adalimumab every two weeks by SC injection.
- IXE80Q2W - Blinded Treatment: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every two weeks by subcutaneous injection.
- IXE80Q4W - Blinded Treatment: Participants received starting dose of either 80 milligrams (mg) or 160mg Ixekizumab at week 0 followed by 80mg Ixekizumab every four weeks by subcutaneous injection.
- ADA/PBO - Washout Treatment Period: Participants received placebo by subcutaneous injection
- PBO/IXE - Extended Treatment Period: Participants received starting dose of 160mg Ixekizumab at week 16 followed by 80mg Q2W or 80mg Q4W by subcutaneous injection.
- ADA/PBO/IXE - Extended Treatment Period: Participants received 80mg Ixekizumab Q2W or 80mg Q4W by subcutaneous injection.
- IXE80Q2W/IXE80Q2W - Extended Treatment: Participants received 80mg Ixekizumab every two weeks by subcutaneous injection.
- IXE80Q4W/IXE80Q4W - Extended Treatment: Participants received 80mg Ixekizumab every four weeks by subcutaneous injection.
- PBO-follow-up Period; IXE80Q2W-follow-up Period; IXE80Q4W-follow-up Period: Participants did not receive any intervention.
Arm/Group | Placebo - Blinded Treatment | Adalimumab 40mg - Blinded Treatment | IXE80Q2W - Blinded Treatment | IXE80Q4W - Blinded Treatment | ADA/PBO - Washout Treatment Period | PBO/IXE - Extended Treatment Period | ADA/PBO/IXE - Extended Treatment Period | IXE80Q2W/IXE80Q2W - Extended Treatment | IXE80Q4W/IXE80Q4W - Extended Treatment | PBO-follow-up Period | IXE80Q2W-follow-up Period | IXE80Q4W-follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/90 | 0/83 | 0/81 | 0/88 | 0/86 | 0/86 | 0/79 | 0/78 | 0/1 | 0/24 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/86 | 3/90 | 1/83 | 1/81 | 0/88 | 4/86 | 7/86 | 3/79 | 4/78 | 0/1 | 0/24 | 0/16
Other Adverse Events (participants affected / at risk) | 12/86 | 16/90 | 18/83 | 11/81 | 8/88 | 26/86 | 20/86 | 21/79 | 14/78 | 1/1 | 2/24 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Blinded Treatment (N=86) | Adalimumab 40mg - Blinded Treatment (N=90) | IXE80Q2W - Blinded Treatment (N=83) | IXE80Q4W - Blinded Treatment (N=81) | ADA/PBO - Washout Treatment Period (N=88) | PBO/IXE - Extended Treatment Period (N=86) | ADA/PBO/IXE - Extended Treatment Period (N=86) | IXE80Q2W/IXE80Q2W - Extended Treatment (N=79) | IXE80Q4W/IXE80Q4W - Extended Treatment (N=78) | PBO-follow-up Period (N=1) | IXE80Q2W-follow-up Period (N=24) | IXE80Q4W-follow-up Period (N=16)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 0/15 (0) | 1/17 (1) | 0/19 (0) | 0/13 (0) | 0/17 (0) | 0/15 (0) | 0/16 (0) | 0/18 (0) | 0/13 (0) | 0 (0) | 0/9 (0) | 0/3 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Blinded Treatment (N=86) | Adalimumab 40mg - Blinded Treatment (N=90) | IXE80Q2W - Blinded Treatment (N=83) | IXE80Q4W - Blinded Treatment (N=81) | ADA/PBO - Washout Treatment Period (N=88) | PBO/IXE - Extended Treatment Period (N=86) | ADA/PBO/IXE - Extended Treatment Period (N=86) | IXE80Q2W/IXE80Q2W - Extended Treatment (N=79) | IXE80Q4W/IXE80Q4W - Extended Treatment (N=78) | PBO-follow-up Period (N=1) | IXE80Q2W-follow-up Period (N=24) | IXE80Q4W-follow-up Period (N=16)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 2 (33) | 3 (6) | 7 (37) | 0 (0) | 0 (0) | 8 (53) | 8 (24) | 6 (34) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (7) | 5 (6) | 6 (6) | 6 (6) | 17 (22) | 7 (8) | 7 (9) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (3) | 4 (4) | 7 (8) | 2 (2) | 4 (4) | 4 (5) | 8 (9) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0/15 (0) | 1/17 (1) | 0/19 (0) | 0/13 (0) | 0/17 (0) | 0/15 (0) | 0/16 (0) | 0/18 (0) | 0/13 (0) | 0 (0) | 0/9 (0) | 0/3 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/15 (0) | 1/17 (1) | 0/19 (0) | 0/13 (0) | 0/17 (0) | 0/15 (0) | 0/16 (0) | 0/18 (0) | 0/13 (0) | 0 (0) | 0/9 (0) | 0/3 (0)
Adnexal torsion (Reproductive system and breast disorders) | 0/15 (0) | 1/17 (1) | 0/19 (0) | 0/13 (0) | 0/17 (0) | 0/15 (0) | 0/16 (0) | 0/18 (0) | 0/13 (0) | 0 (0) | 0/9 (0) | 0/3 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0/15 (0) | 0/17 (0) | 0/19 (0) | 0/13 (0) | 0/17 (0) | 0/15 (0) | 0/16 (0) | 0/18 (0) | 0/13 (0) | 1 (1) | 0/9 (0) | 0/3 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1/15 (1) | 0/17 (0) | 0/19 (0) | 0/13 (0) | 0/17 (0) | 0/15 (0) | 0/16 (0) | 0/18 (0) | 0/13 (0) | 0 (0) | 0/9 (0) | 0/3 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-12-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT02696785/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT02696785/SAP_001.pdf